CLINICAL TRIAL: NCT00938600
Title: Antenatal Vitamin D Supplementation to Improve Neonatal Health Outcomes in Dhaka, Bangladesh: Preliminary Dose-finding and Safety Study
Brief Title: Antenatal Vitamin D3 Dose-finding and Safety Study
Acronym: AViDD-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Abdullah Baqui, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHU-1819
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy; Nutritional Status; Vitamin D
Keywords: pharmacokinetics; safety
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A1 - non-pregnant single-dose (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- A2 - non-pregnant; weekly dose (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- B1 - pregnant; single-dose (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- B2 - pregnant; weekly dose (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- C1 - active control; pregnant women (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 oral liquid 70,000 IU once
  Other Names: Cholecalciferol; Vigantol Oil
  Arms: A1 - non-pregnant single-dose; B1 - pregnant; single-dose
Dietary Supplement: Vitamin D3 — Vitamin D3 oral liquid 70,000 IU as loading dose, then 35,000 IU weekly thereafter for 10 weeks (non-pregnant) or until delivery (pregnant)
  Other Names: Cholecalciferol; Vigantol Oil
  Arms: A2 - non-pregnant; weekly dose; B2 - pregnant; weekly dose
Dietary Supplement: Vitamin D3 — Vitamin D3 14,000 IU per week by mouth, starting at 27-30 weeks gestation and continued until delivery.
  Other Names: Cholecalciferol; Vigantol Oil
  Arms: C1 - active control; pregnant women

SUMMARY:
This is a preliminary study of oral vitamin D3 supplementation in pregnant and non-pregnant women of reproductive age in Bangladesh. The primary objective of the study is to identify a dose of vitamin D3 that can safely be administered during pregnancy to improve the vitamin D status of the mother and infant.

DETAILED DESCRIPTION:
Vitamin D deficiency is common among pregnant and non-pregnant Bangladeshi women. The consequences of vitamin D deficiency during pregnancy are unknown, but increasing evidence suggests it may compromise fetal growth and development of the immune system. We hypothesize that vitamin D deficiency in pregnant women has an adverse effect on the newborn's defenses against infectious diseases in early infancy, and thus contributes to the high rates of neonatal mortality in South Asia. Randomized controlled trials of antenatal vitamin D supplementation are needed to test this hypothesis. However, preliminary studies are first necessary to establish a safe and efficacious dose of vitamin D to be used in such trials. In the proposed study, we will measure the response of the 25-hydroxyvitamin D serum concentration (a biomarker of vitamin D status) to oral vitamin D3 supplementation in pregnant women and non-pregnant women of reproductive age. The goal is to establish a safe, efficacious and feasible weekly vitamin D supplementation regimen for use in future trials. Five groups of approximately 15 women (3 groups of pregnant and 2 groups of non-pregnant women; total up to 75 women) will be supplemented and followed closely for 10 weeks (non-pregnant women) or until delivery (pregnant participants). The primary outcomes will be the change in 25-hydroxyvitamin D concentrations following vitamin D supplementation, and safety parameters that reflect calcium regulation (serum albumin-adjusted calcium concentrations and urine calcium excretion) and fetal development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, age 18 to < 35 years, who are clients at the Shimantik clinic or friends/relatives of Shimantik clients.
* Current permanent residence in Dhaka at a fixed address, and have plans to stay in Dhaka for at least 4 months.
* Pregnant women: Enrolled between 26th and 30th week of gestation (participants enrolled in 26th week will not start on-study until the 27th week or later), with a normal medical and obstetric history. Gestational age will be estimated based on the first day of the last menstrual period (LMP).
* Informed consent provided after having an opportunity to consult with husband and/or family members.

Exclusion Criteria:

* Current self-reported use of any non-food-based dietary supplements containing vitamin D (i.e., commercial micronutrient pills or capsules containing vitamin D).
* Current use of anti-convulsant or anti-mycobacterial (tuberculosis) medications.
* Severe anemia (hemoglobin concentration < 70 g/L).
* Hypertension (systolic blood pressure >= 140 mmHg or diastolic blood pressure >= 90 mmHg on at least two measurements).
* In pregnant women: previous history of giving birth to an infant with congenital anomalies.
* In non-pregnant women: currently breast-feeding.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D concentration | 6 scheduled timepoints during supplementation period
Serum calcium concentration (albumin-corrected) | 6 scheduled timepoints during supplementation period
Urine calcium: creatinine ratio | 7-8 scheduled timepoints during supplementation period

SECONDARY OUTCOMES:
Blood pressure | Weekly during supplementation period
Urinary protein excretion | Weekly during supplementation period
Maternal weight | Weekly during supplementation period
Birth anthropometry | At birth
Neonatal echocardiography | Neonatal period
Fetal LL-37 expression/secretion in saliva, vernix, and cord tissue | Birth

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Baqui, MBBS, Principal Investigator — The Johns Hopkins Bloomberg School of Public Health; Rubhana Raqib, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Shams El Arifeen, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Daniel E Roth, MD, Study Director — The Johns Hopkins Bloomberg School of Public Health
Locations (1):
- SHIMANTIK Maternity Centre, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Background] Islam MZ, Shamim AA, Kemi V, Nevanlinna A, Akhtaruzzaman M, Laaksonen M, Jehan AH, Jahan K, Khan HU, Lamberg-Allardt C. Vitamin D deficiency and low bone status in adult female garment factory workers in Bangladesh. Br J Nutr. 2008 Jun;99(6):1322-9. doi: 10.1017/S0007114508894445. PMID 18430266
- [Background] Islam MZ, Lamberg-Allardt C, Karkkainen M, Outila T, Salamatullah Q, Shamim AA. Vitamin D deficiency: a concern in premenopausal Bangladeshi women of two socio-economic groups in rural and urban region. Eur J Clin Nutr. 2002 Jan;56(1):51-6. doi: 10.1038/sj.ejcn.1601284. PMID 11840180
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Roth DE, Al Mahmud A, Raqib R, Black RE, Baqui AH. Pharmacokinetics of a single oral dose of vitamin D3 (70,000 IU) in pregnant and non-pregnant women. Nutr J. 2012 Dec 27;11:114. doi: 10.1186/1475-2891-11-114. PMID 23268736